CLINICAL TRIAL: NCT03591770
Title: The Immunogenicity and Safety of Shingrix Vaccine in Patients With Moderate to Severe Ulcerative Colitis on Tofacitinib
Brief Title: Shingrix Vaccine in Patients With Moderate to Severe Ulcerative Colitis on Tofacitinib
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit adequate numbers of participants to answer the research question.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-37673
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Shingrix vaccine; tofacitinib monotherapy; anti-TNF monotherapy; anti-TNF agent; thiopurine; aminosalicylates
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- UC patients on tofacitinib monotherapy (Experimental): Ulcerative Colitis patients on Tofacitinib monotherapy, all patients will be treated with the standard Tofacitinib and will receive Shingrix vaccine.
  Interventions: Biological: SHINGRIX
- UC patients on anti-TNF monotherapy (Active Comparator): Ulcerative Colitis patients on anti-TNF monotherapy, all patients will be treated with the standard anti-TNF monotherapy (adalimumab, golimumab, certolizumab, infliximab)and will receive Shingrix vaccine.
  Interventions: Biological: SHINGRIX
- UC patients on anti-TNF and a thiopurine (Active Comparator): Ulcerative Colitis patients on anti-TNF and a thiopurine, all patients will be treated with the standard anti-TNF monotherapy (adalimumab, golimumab, certolizumab, infliximab) and thiopurine (6-mercaptopurine, azathioprine) and will receive Shingrix vaccine.
  Interventions: Biological: SHINGRIX
- UC pts. on aminosalicylates or off immunomodulatory therapy (Active Comparator): Ulcerative Colitis patients on non-immunosuppressive therapy or 5-aminosalicylates, all patients will be treated with the standard non-immunosuppressive therapy or 5-aminosalicylates and will receive Shingrix vaccine.
  Interventions: Biological: SHINGRIX

INTERVENTIONS:
Biological: SHINGRIX — SHINGRIX is a vaccine indicated for prevention of herpes zoster (shingles) in adults aged 50 years and older.
  SHINGRIX is a suspension for injection supplied as a single-dose vial of lyophilized gE antigen component to be reconstituted with the accompanying vial of AS01B adjuvant suspension component. A single dose after reconstitution is 0.5 mL.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
  Other Names: Recombinant zoster vaccine

SUMMARY:
Patients with ulcerative colitis (UC), a chronic inflammatory bowel disease (IBD), have been shown to be at increased risk of developing certain infections, such as shingles from the Herpes Zoster (HZ) virus, as a result of their underlying disease. Patients with UC are also often treated with immunosuppressants, and research has shown that IBD patients on immunosuppressants have an impaired immune response to vaccination in comparison to immunocompetent controls. Because UC patients are often treated with immunosuppressants, the live HZ vaccine was not recommended in these patients. Shingrix, however, is a new inactivated vaccine recently approved by the FDA for prevention of HZ in adults age 50 and older, and Shingrix should be safe to administer in IBD patients because it does not contain live HZ virus. Data on efficacy of the Shingrix vaccine also appears promising in immunocompromised patients.

Tofacitinib citrate (Xeljanz), an immunosuppressant that works by inhibiting the Janus kinase pathway, is currently approved for treatment of certain inflammatory diseases such as rheumatoid arthritis and psoriasis. The drug is currently awaiting FDA-approval for use in moderate-to-severe UC but has been used off-label in various settings. Notably, tofacitinib was associated with an increased risk of HZ in patients with rheumatoid arthritis and psoriasis.

The research hypothesis is that UC patients on tofacitinib will mount an adequate response and that the response will be slightly diminished compared to non-immunosuppressed IBD patients, comparable to those on anti-tumor necrosis alpha (anti-TNF) monotherapy, and superior to those on anti-TNF therapy in combination with a thiopurine. Strong cell mediated immunity is shown to prevent reactivation of HZ, and demonstrating a robust immune response to Shingrix may serve as a surrogate for a reduced risk of developing shingles and might alleviate prescribers' concerns regarding the use of tofacitinib. The results will also serve as pilot data to inform larger future studies evaluating the actual risk of developing shingles in patients on tofacitinib who receive Shingrix.

DETAILED DESCRIPTION:
The purpose of this study is to determine the immune response from the new Shingrix vaccine in UC patients on tofacitinib monotherapy in comparison to other UC therapies. the investigators plan to determine this by vaccinating IBD patients on (a) tofacitinib monotherapy, (b) anti-TNF monotherapy, (c) anti-TNF combination therapy with a thiopurine, or (d) aminosalicylates or other non-immunosuppressive therapy with the new Shingrix vaccine and measuring markers of cell-mediated immunity before vaccination and at one and six months after the last vaccine dose. Cell-mediated immunity will be measured with an interferon gamma (IFNγ) enzyme linked immunospot (ELISPOT) test to assess T-cell response. Humoral immunity will also be measured with an enzyme-linked immunosorbent assay (ELISA) kit to quantify antibody concentrations of Varicella Zoster Virus (VZV), the pathogen that when reactivated results in shingles.

The study population will include adult patients aged 50 or older with UC (diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria) receiving care at Boston Medical Center, Hospital of the University of Pennsylvania, or University of Wisconsin Hospital and Clinics. There is no randomization or use of placebo in this study. Four study groups (each containing 25 subjects) will be established -- 1. Group A - UC patients on tofacitinib monotherapy. 2. Group B - UC patients receiving anti-TNF monotherapy (adalimumab, golimumab, infliximab). 3. Group C - UC patients on an anti-TNF agent and a thiopurine (6-mercaptopurine, azathioprine). Group D - UC patients on non-immunosuppressive therapy or 5-aminosalicylates. For each subject, 3 total samples will be collected.

Methods: Eligible patients with UC will be recruited from the Center for Digestive Diseases at Boston Medical Center, the Hospital of the University of Pennsylvania, or the University of Wisconsin Hospital and Clinics. Patients will be screened for participation in the study and recruited by their primary gastroenterologist. In clinic, a handout of the risks and benefits of the clinically indicated vaccine (Shingrix) will be given to each patient from their primary gastroenterologist for their review. Patients will have the opportunity to opt in or out of the study early in the consent process upon review of the handout. If a patient elects to participate in the study, patients will sign the consent, be entered into the study with assignment of a Subject ID number, and complete the initial study assessments:

Subject contacts:

* 1 - Baseline/Enrollment Visit 1 (Day 0): Subjects will have a comprehensive medical history and physical exam performed, including vaccination history and all medications over past 30 days. They will also complete a Simple Clinical Colitis Activity Index (SCCAI) questionnaire. A baseline blood sample of approximately 20mL (4 tablespoons) will then be obtained. If proof of past varicella infection is met by appropriate history, subjects will receive the Shingrix vaccine indicated based on their vaccination history as recommended by their gastroenterologist; otherwise subjects will follow-up in 1 week to review confirmatory serology results and receive vaccine if indicated. The Shingrix vaccine will be given in a two-dose series (0.5 mL each) administered intramuscularly -first dose at Month 0 followed by a second dose anytime between 2 and 6 months later. Subjects will be instructed to call the study team for any concerns or any development of fever, chills, rash or other concerning symptom.
* 2- Follow up Visit 2 (approximately day 7): This visit is only needed for patients who require serologic confirmation of past varicella infection, therefore patients who meet proof for past varicella infection by appropriate history do not require serologic confirmation and will NOT be scheduled for this visit. Subjects will review results of the VZV antibody level test with their provider. If VZV antibody levels are positive, subjects will receive the Shingrix vaccine indicated based on their vaccination history as recommended by their gastroenterologist. Subjects will be instructed to call the study team for any concerns or any development of fever, chills, rash or other concerning symptom.
* 3 - Follow up Phone Call 1 (approximately day 14): Subjects will receive a follow-up phone call to identify any adverse effects including fevers or chills, rash, and visits to the emergency room or to their primary care physicians. They will also be reminded about their follow up visit.
* 4 - Follow up Visit 3 (approximately day 60): Subjects will complete a SCCAI questionnaire, and information will be collected to identify any adverse effects including fevers or chills, rash, and visits to the emergency room or to their primary care physician. The 2nd dose of the Shingrix vaccine will be administered.
* 5 - Follow up Phone Call 2 (approximately day 72): Subjects will receive a follow-up phone call to identify any adverse effects including fevers or chills, rash, and visits to the emergency room or to their primary care physicians. They will also be reminded about their follow up visit.
* 6 - Follow up Visit 4 (approximately day 90): Subjects will complete a SCCAI questionnaire, and information will be collected to identify any adverse effects including fevers or chills, rash, and visits to the emergency room or to their primary care physician. A blood sample of approximately 20mL (4 tablespoons) will then be obtained.
* 7 - Follow up Visit 5 (approximately day 240): Subjects will complete a SCCAI questionnaire, and information will be collected to identify any adverse effects including fevers or chills, rash, and visits to the emergency room or to their primary care physician. A blood sample of approximately 20mL (4 tablespoons) will then be obtained.

The entire procedure will be identically performed at the additional sites outside of Boston Medical Center. Subjects' duration of participation will range from 8 to 12 months, depending on when the 2nd vaccine dose is administered.

ELIGIBILITY:
Inclusion Criteria:

1. Proof of primary varicella infection (chicken pox) either by appropriate history (as defined by ACIP) or otherwise confirmed with a positive VZV IgG antibody level
2. Patient has a history of ulcerative colitis (UC) diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria
3. Patient is receiving one of the following treatments for their UC:

Group A: Tofacitinib monotherapy, Group B: Anti-TNF monotherapy (adalimumab, golimumab, certolizumab pegol, infliximab), Group C: Anti-TNF combination therapy with a thiopurine (6 mercaptopurine, azathioprine), Group D: 5-aminosalicylates or other non-immunomodulatory therapy.

Exclusion Criteria:

1. Previous receipt of any HZ vaccine
2. Allergy to zoster vaccine or a component of the vaccine
3. Other underlying chronic medical conditions that could affect immunogenicity to vaccines (rheumatoid arthritis, psoriasis etc.)
4. History of herpes zoster infection or post herpetic neuralgia
5. Patient cannot or will not provide written informed consent
6. Patient is on a non-licensed or experimental immunomodulator
7. Patient is on methotrexate
8. Patient has received immunoglobulin therapy or blood products with the past month
9. Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharmeel K Wasan, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated before any participants were assigned to the arm on anti-TNF and thiopurine.
Groups:
- UC Patients on Anti-TNF Monotherapy: Ulcerative Colitis patients on anti-TNF monotherapy, all patients will be treated with the standard anti-TNF monotherapy and will receive Shingrix vaccine.
- UC Patients on Anti-TNF and a Thiopurine: Ulcerative Colitis patients on anti-TNF and a thiopurine, all patients will be treated with the standard anti-TNF monotherapy and thiopurine (6-mercaptopurine, azathioprine) and will receive Shingrix vaccine.
Period: Overall Study
Arm/Group | UC Patients on Tofacitinib Monotherapy | UC Patients on Anti-TNF Monotherapy | UC Patients on Anti-TNF and a Thiopurine | UC Pts. on Aminosalicylates or Off Immunomodulatory Therapy
Started | 3 | 8 | 0 | 4
Completed | 1 | 0 | 0 | 0
Not Completed | 2 | 8 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The study was terminated before any participants were assigned to the arm on anti-TNF and thiopurine.
Groups:
- Total: Total of all reporting groups
Arm/Group | UC Patients on Tofacitinib Monotherapy | UC Patients on Anti-TNF Monotherapy | UC Patients on Anti-TNF and a Thiopurine | UC Pts. on Aminosalicylates or Off Immunomodulatory Therapy | Total
Number analyzed (Participants) | 3 | 8 | 0 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (7) | 54 (10) |  | 58 (6) | 51 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 |  | 3 | 9
  Male | 3 | 2 |  | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 |  | 1 | 6
  Not Hispanic or Latino | 2 | 4 |  | 3 | 9
  Unknown or Not Reported | 0 | 0 |  | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or Af Am | 0 | 2 |  | 1 | 3
  White | 2 | 2 |  | 2 | 6
  Unk or Not reported | 1 | 4 |  | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 3 | 8 |  | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in the Immunogenicity of the Herpes Zoster Subunit Vaccine in UC Patients
Description: Immunogenicity will be assessed by the change in cell mediated immunity (CMI) as measured by ELISPOT from pre-immunization to 1 month after receiving second dose of booster vaccine post-immunization. ELISPOT is an enzyme-linked assay for detecting and enumerating cytokine-producing lymphocytes. A colored spot indicates a cell producing IFNγ. Each well will be inspected and cytokine-producing cells will be counted using AID® imaging system. Any well with more than 300 spots will be considered too numerous to count and reported as >300 cells/well. It will be measured from pre-immunization to 1 month after receiving second dose of booster vaccine post-immunization.
Time Frame: Baseline and approximately 90 days
Population: The study was terminated before any participants were assigned to the arm on anti-TNF and thiopurine so there are no participants enrolled in this arm. For the other three arms there were not enough participants enrolled to test the samples for this outcome measure as the minimum number needed for this test is 25. Therefore, there are no data for this outcome measure.
Arm/Group | UC Patients on Tofacitinib Monotherapy | UC Patients on Anti-TNF Monotherapy | UC Patients on Anti-TNF and a Thiopurine | UC Pts. on Aminosalicylates or Off Immunomodulatory Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: The Number of Participants With Vaccine Adverse Effects at 1 Month
Description: Vaccine adverse effects will be documented following immunization by evaluating participants at each clinic visit and from a phone call by study personnel.
Time Frame: 1 month
Population: The study was terminated before any participants were assigned to the arm on anti-TNF and thiopurine so there are no participants enrolled in this arm.
Measure: Count of Participants; unit: Participants
Groups:
- UC Patients on Tofacitinib Monotherapy: Ulcerative Colitis patients on Tofacitinib monotherapy, all patients will be treated with the standard Tofacitinib and will receive Shingrix vaccine.
  SHINGRIX: SHINGRIX is a vaccine indicated for prevention of herpes zoster (shingles) in adults aged 50 years and older.
  SHINGRIX is a suspension for injection supplied as a single-dose vial of lyophilized gE antigen component to be reconstituted with the accompanying vial of AS01B adjuvant suspension component. A single dose after reconstitution is 0.5 mL.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
- UC Patients on Anti-TNF Monotherapy: Ulcerative Colitis patients on anti-TNF monotherapy, all patients will be treated with the standard anti-TNF monotherapy (adalimumab, golimumab, certolizumab, infliximab)and will receive Shingrix vaccine.
  SHINGRIX: SHINGRIX is a vaccine indicated for prevention of herpes zoster (shingles) in adults aged 50 years and older.
  SHINGRIX is a suspension for injection supplied as a single-dose vial of lyophilized gE antigen component to be reconstituted with the accompanying vial of AS01B adjuvant suspension component. A single dose after reconstitution is 0.5 mL.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
- UC Patients on Anti-TNF and a Thiopurine: Ulcerative Colitis patients on anti-TNF and a thiopurine, all patients will be treated with the standard anti-TNF monotherapy (adalimumab, golimumab, certolizumab, infliximab) and thiopurine (6-mercaptopurine, azathioprine) and will receive Shingrix vaccine.
  SHINGRIX: SHINGRIX is a vaccine indicated for prevention of herpes zoster (shingles) in adults aged 50 years and older.
  SHINGRIX is a suspension for injection supplied as a single-dose vial of lyophilized gE antigen component to be reconstituted with the accompanying vial of AS01B adjuvant suspension component. A single dose after reconstitution is 0.5 mL.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
- UC Pts. on Aminosalicylates or Off Immunomodulatory Therapy: Ulcerative Colitis patients on non-immunosuppressive therapy or 5-aminosalicylates, all patients will be treated with the standard non-immunosuppressive therapy or 5-aminosalicylates and will receive Shingrix vaccine.
  SHINGRIX: SHINGRIX is a vaccine indicated for prevention of herpes zoster (shingles) in adults aged 50 years and older.
  SHINGRIX is a suspension for injection supplied as a single-dose vial of lyophilized gE antigen component to be reconstituted with the accompanying vial of AS01B adjuvant suspension component. A single dose after reconstitution is 0.5 mL.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
Arm/Group | UC Patients on Tofacitinib Monotherapy | UC Patients on Anti-TNF Monotherapy | UC Patients on Anti-TNF and a Thiopurine | UC Pts. on Aminosalicylates or Off Immunomodulatory Therapy
Number analyzed (Participants) | 3 | 8 | 0 | 4
Participants | 0 | 0 |  | 0

3. Secondary Outcome: Number of Participants With Vaccine Adverse Effects at 8 Months (6 Months Post-immunization)
Description: as for outcome 2
Time Frame: 8 months (6 months post-immunization)
Population: The study was terminated before any participants were assigned to the arm on anti-TNF and thiopurine so there are no participants enrolled in this arm. At 8 months, all participants in the other 3 arms, except for one in the UC patients on tofacitinib monotherapy, were lost to follow-up so there are no data for the UC patients on anti-TNF monotherapy and the UC pts. on aminosalicylates or off immunomodulatory therapy arms.
Measure: Count of Participants; unit: Participants
Arm/Group | UC Patients on Tofacitinib Monotherapy | UC Patients on Anti-TNF Monotherapy | UC Patients on Anti-TNF and a Thiopurine | UC Pts. on Aminosalicylates or Off Immunomodulatory Therapy
Number analyzed (Participants) | 1 | 0 | 0 | 0
Participants | 0 |  |  |

4. Secondary Outcome: Number of Participants Classified by Disease Activity
Description: The Simple Clinical Colitis Activity Index (SCCAI) will be used to measure disease activity. It is a questionnaire with six subscore topics with scores defined by UC signs and symptoms from 0 to 4 for a range of scores from 0 to 17. Total scores are interpreted as: Remission = score of 0 to 4 points, Mild Activity = score of 5 to 7 points, Moderate Activity = Score of 8 to 16 points, and Severe Activity = Score of > 16 points.
Time Frame: Baseline, 2 months, and 8 months (6 months post-immunization)
Population: 1. The study was terminated before any participants were assigned to the arm on anti-TNF and thiopurine so there are no participants enrolled in this arm.
  2. None of the participants in the arm on UC pts. on aminosalicylates or off immunomodulatory therapy completed any of the questionnaires for any of the time frames, so there are no data for this arm.
Measure: Count of Participants; unit: Participants
Arm/Group | UC Patients on Tofacitinib Monotherapy | UC Patients on Anti-TNF Monotherapy | UC Patients on Anti-TNF and a Thiopurine | UC Pts. on Aminosalicylates or Off Immunomodulatory Therapy
Number analyzed (Participants) | 3 | 3 | 0 | 0
Participants
  Baseline: Remission | 2 | 1 |  |
  Baseline: Mild Activity | 1 | 1 |  |
  Baseline: ModerateActivity | 0 | 1 |  |
  Baseline: Severe Activity | 0 | 0 |  |
  2 months: number analyzed (Participants) | 2 | 3 | 0 | 0
  2 months: Remission | 2 | 2 |  |
  2 months: Mild Activity | 0 | 0 |  |
  2 months: ModerateActivity | 0 | 1 |  |
  2 months: Severe Activity | 0 | 0 |  |
  8 months: number analyzed (Participants) | 1 | 0 | 0 | 0
  8 months: Remission | 1 |  |  |
  8 months: Mild Activity | 0 |  |  |
  8 months: ModerateActivity | 0 |  |  |
  8 months: Severe Activity | 0 |  |  |

ADVERSE EVENTS:
Time Frame: about 8 months
Description: There were no participants assigned to the group with UC patients on anti TNF and thiopurine.
Arm/Group | UC Patients on Tofacitinib Monotherapy | UC Patients on Anti-TNF Monotherapy | UC Patients on Anti-TNF and a Thiopurine | UC Pts. on Aminosalicylates or Off Immunomodulatory Therapy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/8 | 0/0 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/8 | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/8 | 0/0 | 0/4

LIMITATIONS AND CAVEATS:
The study was halted since the investigators were unable to recruit adequate numbers of participants to answer the research question. There were no patients enrolled in the anti-TNF and a thiopurine group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT03591770/Prot_SAP_000.pdf